CLINICAL TRIAL: NCT05739383
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Effect of Inclisiran on Preventing Major Adverse Cardiovascular Events in High-risk Primary Prevention Patients (VICTORION-1 PREVENT)
Brief Title: A Study of Inclisiran to Prevent Cardiovascular Events in High-risk Primary Prevention Patients.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CKJX839D12302
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary Prevention of Atherosclerotic Cardiovascular Disease
Keywords: Inclisiran; PCSK9; primary prevention; cardiovascular disease; MACE; myocardial infarction; stroke; LDL-C; hyperlipidemia; hypercholesterolemia; dyslipidemia; cholesterol; Coronary Artery Disease (CAD); Non-Obstructive Coronary Artery Disease (NOCAD); Coronary Artery Calcium; Coronary artery stenosis; Coronary angiogram
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Hyperlipidemias; Hypercholesterolemia; Dyslipidemias; Coronary Artery Disease; Coronary Stenosis | interventions — ALN-PCS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran sodium 300mg (Experimental): Inclisiran sodium 300 mg in 1.5 mL solution for injection (subcutaneous) in pre-filled syringe.
  Randomized in a 1:1 ratio with matching placebo
  Interventions: Drug: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL
- Placebo (Placebo Comparator): Matching placebo in 1.5ml pre-filled syringe. Randomized in a 1:1 ratio with Inclisiran.
  Interventions: Drug: Placebo in 1.5ml

INTERVENTIONS:
Drug: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL — Subcutaneous injection in pre-filled syringe.
  Other Names: KJX839
  Arms: Inclisiran sodium 300mg
Drug: Placebo in 1.5ml — Matching placebo in 1.5ml solution for injection
  Arms: Placebo

SUMMARY:
CKJX839D12302 is a pivotal Phase III study designed to test the hypothesis that treatment with inclisiran sodium 300 milligram (mg) subcutaneous (s.c.) administered on Day 1, Day 90, and every 6 months thereafter in patients at high cardiovascular (CV) risk without a prior major atherosclerotic cardiovascular disease (ASCVD) event will significantly reduce the risk of 4-Point-Major Adverse Cardiovascular Events (4P-MACE) defined as a composite of CV death, non-fatal myocardial infarction (MI), non-fatal ischemic stroke, and urgent coronary revascularization, compared to placebo.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate inclisiran sodium 300 mg s.c. (equivalent to 284 mg inclisiran) compared to placebo on reducing the risk of 4P-MACE in adult patients at high risk for their first major adverse cardiovascular event.

Randomized participants will receive study medication (inclisiran or placebo), administered s.c. on Day 1, Day 90, then every 6 months thereafter. This is an event-driven study. Therefore, the study will continue until the required number of clinical events have occurred across both treatment arms, and all participants have a minimum of 3 years of follow-up during the double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* At an increased risk for a first MACE (i.e., no prior major ASCVD event), defined as any one of the following:

  1. Evidence of atherosclerotic coronary artery disease (CAD) on computer tomography (CT) or invasive coronary angiogram defined as a coronary artery stenosis ≥20% but <50% in the left main coronary artery or stenosis ≥20% but <70% in any other major epicardial coronary artery, or
  2. Coronary artery calcium (CAC) score obtained by CT-scan ≥100 Agatston units, or
  3. High 10-year ASCVD risk ≥20%, or
  4. Intermediate 10-year ASCVD risk 7.5% - <20% with at least 2 risk-enhancing factors.
* LDL-C ≥70 mg/dL (≥1.81 mmol/L) but <190 mg/dL (<4.91 mmol/L) at the screening visit. If on a background lipid lowering therapy, the dose should be stable for at least 4 weeks prior to the screening visit and the participant should be willing to remain on this background therapy for the entire duration of the study.

Exclusion Criteria:

* History of major ASCVD event.
* History of, or planned, ischemia-driven revascularization in a coronary or extracoronary arterial bed prior to randomization
* Absence of coronary atherosclerosis on a CT angiogram or an invasive coronary angiogram in the 2 years prior to randomization
* Coronary artery calcium (CAC) score of 0 obtained in the 2 years prior to randomization
* Active liver disease or hepatic dysfunction
* Previous, current, or planned treatment with a monoclonal antibody (mAb) directed toward proprotein convertase subtilisin/kexin type 9 (PCSK9) (e.g., evolocumab, alirocumab)
* Pregnant or nursing (lactating) women
* Women of childbearing potential unless they are using effective methods of contraception while taking study treatment which includes for 6 months after last study drug administration

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14082 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2029-04-16 (Estimated); Study Completion 2029-04-16 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of 4P-MACE | Time to the first occurrence of 4P-MACE (up to approximately 75 months)
  4-Point-Major Adverse Cardiovascular Events (4P-MACE): composite of cardiovascular death, non-fatal myocardial infarction, non-fatal ischemic stroke, and urgent coronary revascularization.

SECONDARY OUTCOMES:
Time to the first occurrence of 3P-MACE | Time to the first occurrence of 3P-MACE (up to approximately 75 months)
  3-Point-Major Adverse Cardiovascular Events (3P-MACE): composite of cardiovascular death, non-fatal myocardial infarction, and non-fatal ischemic stroke)
Total number of first or repeated CV events (4P MACE) | up to 75 months
  Total 4P-MACE (composite of cardiovascular death, non-fatal myocardial infarction, non-fatal ischemic stroke, and urgent coronary revascularization)
Total number of first or repeated CV events (3P MACE) | up to 75 months
  Total 3P-MACE (composite of cardiovascular death, non-fatal myocardial infarction, and non-fatal ischemic stroke)
Time to occurrence of Cardiovascular death | Time to Cardiovascular death (up to 75 months)
  CV death is defined as death due to cardiovascular events.
Time to occurrence of death due to any reason | Time to all-cause mortality (up to 75 months)
  All-cause mortality is death due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (836):
- United States (245):
  - Central Alabama Research, Birmingham, Alabama
  - UAB St Vincents, Birmingham, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - G and L Research LLC, Foley, Alabama
  - Longwood Research, Huntsville, Alabama
  - CB Flock Corporation, Mobile, Alabama
  - Mobile Heart Specialists, Mobile, Alabama
  - The Center for Clinical Trials, Saraland, Alabama
  - Alaska Heart and Vascular, Anchorage, Alaska
  - Synexus, Glendale, Arizona
  - Lenzmeier Family Practice, Glendale, Arizona
  - Avacare Center for Dermatology, Phoenix, Arizona
  - Clinical Research Inst of Arizona, Sun City West, Arizona
  - Clinical Research Advantage Fiel Family and Sports Med, PC, Tempe, Arizona
  - Synexus Clinical Research US Inc, Tucson, Arizona
  - Cardiovascular Res Found, Beverly Hills, California
  - National Heart Institute, Beverly Hills, California
  - Alliance Clinical, Canoga Park, California
  - Inland Psychiatric Medical Group, Chino, California
  - Valley Clinical Trials Inc, Covina, California
  - Keck Medical Center USC, Los Angeles, California
  - Charles R Drew University of Medicine and Science, Los Angeles, California
  - C for Endo Diabetes and MD, Newhall, California
  - California Medical Research Associates Inc, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Stanford University Medical Center, Palo Alto, California
  - Clinical Trials Research Sacramento, Sacramento, California
  - Cordova Clinical Research, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente San Diego, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Harbor UCLA Medical Center, Torrance, California
  - Cardiology Associates Medical Group, Ventura, California
  - Blue Coast Research Center LLC, Vista, California
  - Interv Cardiology Med Grp, West Hills, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Cardiology Ass of Fairfield County, Stamford, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Nova Clinical Research LLC, Bradenton, Florida
  - Bay Care Medical Group, Clearwater, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Cardiology Research Associates, Daytona Beach, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Personal Physicians Care, Delray Beach, Florida
  - Fleming Island Ctr Clinical Res., Fleming Island, Florida
  - Proactive Clinical Research, Fort Lauderdale, Florida
  - Qway Research, Hialeah, Florida
  - Indago Research and Health Ctr Inc, Hialeah, Florida
  - Sister Life Research Inc, Hialeah, Florida
  - Center for Diabetes and Endocrine Care, Hollywood, Florida
  - South Florida Rsrch Solutions LLC, Hollywood, Florida
  - Zenith Clinical Research, Hollywood, Florida
  - Encore Medical Research, Hollywood, Florida
  - UF Health Science Center, Jacksonville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Infinite Clinical Research, Miami, Florida
  - Springs Medical And Research, Miami, Florida
  - L and C Professional Medical Institute, Miami, Florida
  - Regenerate Clinical Trial, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - A&A Research Group Inc, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - RM Medical Research Inc, Miami Lakes, Florida
  - Eminat Research Group, Miramar, Florida
  - Advent Health Orlando, Orlando, Florida
  - CTMD Research, Palm Springs, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Fam Medical Specialists Of Fl Plc, Plant City, Florida
  - St Johns Center, Ponte Vedra, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - East Coast Inst for Research LLC, Saint Augustine, Florida
  - Cardiovascular Center Of Sarasota, Sarasota, Florida
  - Advanced Medical Research Center, St. Petersburg, Florida
  - James A Haley Veterans Hospital, Tampa, Florida
  - BayCare Health System, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - East Coast Research, Canton, Georgia
  - Javara Research, Fayetteville, Georgia
  - The Jones Center For Diabetes And Endocrine Wellness, Macon, Georgia
  - Atlanta Heart Specialists LLC, Tucker, Georgia
  - East West Research Institute, Honolulu, Hawaii
  - Kootenai Heart Clinic-Sandpoint, Sandpoint, Idaho
  - Endeavor Health Clinical Op- NCH, Arlington Heights, Illinois
  - Chicago Clinical Research Inst, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Flourish Research, Grandwood Park, Illinois
  - Cardiovascular Services, Peoria, Illinois
  - Beacon Health System, Elkhart, Indiana
  - Franciscan Health Services Research Center, Indianapolis, Indiana
  - Buynak Clinical Research PC, Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Cotton O Neil Clinical Res Center, Topeka, Kansas
  - Kansas Heart Hospital, Wichita, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - The Research Group, Lexington, Kentucky
  - Research Integrity LLC, Owensboro, Kentucky
  - Cardiovascular Associates Research, Covington, Louisiana
  - Louisiana Heart Center Research, Covington, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - North Shore Heart and Vascular, Mandeville, Louisiana
  - Bethesda Medical Clinic, Marrero, Louisiana
  - NOLA Care Clinical Research, Metairie, Louisiana
  - Omega Clinical Research, Metairie, Louisiana
  - CV Ins of the South, Opelousas, Louisiana
  - Cardiovascular Solutions LLC, Shreveport, Louisiana
  - Louisiana Heart Center Research, Slidell, Louisiana
  - Monroe Research Llc, West Monroe, Louisiana
  - Southern Clinical Research, Zachary, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants Llc, Beltsville, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - MGH, Boston, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - AA Medical Research Center, Flint, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Central Michigan University, Saginaw, Michigan
  - Troy Internal Medicine Research, Troy, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Essentia Health, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Synexus Clinical Research US Inc, Richfield, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Fairview Health Services, Saint Paul, Minnesota
  - Elite Clinical Research LLC, Jackson, Mississippi
  - Jackson Heart Clinic, Jackson, Mississippi
  - VAMC Research-G V Sonny Montgomery Clinic, Jackson, Mississippi
  - David M Headley Clinic, Port Gibson, Mississippi
  - Cardiology Associates of North MS, Tupelo, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Barnes Jewish Hosp-Washington Univ, St Louis, Missouri
  - St Louis V A Medical Center, St Louis, Missouri
  - St Louis Heart and Vascular, St Louis, Missouri
  - Synexus Clinical Research US Inc, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Lincoln Internal Medicine Associates, Lincoln, Nebraska
  - University of Nebraska Med Center, Omaha, Nebraska
  - Las Vegas Endocrinology, Henderson, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Cardiovas Assoc of Delaware Valley, Elmer, New Jersey
  - New Jersey Heart, Linden, New Jersey
  - Albany Medical College, Albany, New York
  - Capital Cardiology Associates, Albany, New York
  - New York Presbyterian Queens, Flushing, New York
  - Mid Hudson Medical Research PLLC, New Windsor, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Rochester Clinical Research, Rochester, New York
  - Clinical Research Advantage, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Great Lakes Medical Research, Westfield, New York
  - Cary Research Group, Cary, North Carolina
  - Moses Cone Hospital, Greensboro, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - IMA Research, Mount Airy, North Carolina
  - Multispecialty Research Ass Of NC, Raleigh, North Carolina
  - Accellacare, Statesville, North Carolina
  - Adv Imaging Prev and Clin Research, Wilmington, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Altru Health Research Dept., Grand Forks, North Dakota
  - Aultman Hospital, Canton, Ohio
  - Synexus Clinical Research US Inc, Cincinnati, Ohio
  - Synexus Clinical Research, Columbus, Ohio
  - Primed Clinical Research, Dayton, Ohio
  - Providence Medical Group, Dayton, Ohio
  - NexGen Research, Lima, Ohio
  - Rama Research LLC, Marion, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research LLC, Oklahoma City, Oklahoma
  - CCT Hatboro Medical Associates, Horsham, Pennsylvania
  - Capital Area Research LLC, Newport, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Frontier Clinical Research LLC, Smithfield, Pennsylvania
  - Care Access, Warwick, Rhode Island
  - Columbia VA Health Care System, Columbia, South Carolina
  - Bon Secours Medical Group, Greenville, South Carolina
  - TRIBE Clinical Research, Greer, South Carolina
  - Trident Cardiology, Ladson, South Carolina
  - Main Street Physicians Care, Little River, South Carolina
  - Care Access Rapid City, Rapid City, South Dakota
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Wellmont CVA Heart Institute, Greenville, Tennessee
  - Apex Cardiology Research Associates of Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - New Phase Research And Development, Knoxville, Tennessee
  - Accellacare, Knoxville, Tennessee
  - Cardiovascular Res of Knoxville LLC, Powell, Tennessee
  - Tennessee Center For Clinical Trials, Tullahoma, Tennessee
  - Pharma Tex Research, Amarillo, Texas
  - Amarillo Heart Clin Rsh Inst, Amarillo, Texas
  - North Hills Medical Research Inc, Bedford, Texas
  - Clinical Research Solution, Cypress, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - SW Family Medicine Associates, Dallas, Texas
  - Doctors Hospital at Renaissance, Edinburg, Texas
  - David Turbay MD PLLC, El Paso, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Primecare Medical Group, Houston, Texas
  - Northwest Houston Cardiology PA, Houston, Texas
  - MedCare Pharma LLC, Houston, Texas
  - Dallas Heart and Vascular Consultants PA, Houston, Texas
  - Texas Cardiology Assocs Of Houston, Kingwood, Texas
  - Epic Clinical Research, Lewisville, Texas
  - East Texas Research Associates Inc., Livingston, Texas
  - Epic Medical Research, Red Oak, Texas
  - Northeast Clinical Research of San Antonio LLC, San Antonio, Texas
  - Consano Clinical Research LLC, Shavano Park, Texas
  - Javara Research, Stephenville, Texas
  - NRG Wellness Center, Sugarland, Texas
  - Northwest Houston Clinical Research PLLC, Tomball, Texas
  - Comprehensive Center, Weslaco, Texas
  - Intermountain Medical Center, Murray, Utah
  - Diabetes And Endocrine Specialists, Sandy City, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Heart Care Associates P C, Hopewell, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Centricity Research Suffolk Fam Med, Suffolk, Virginia
  - MultiCare Ins Research Innovation, Puyallup, Washington
  - Universal Research Group LLC, Tacoma, Washington
  - Confluence Health Hospital, Wenatchee, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Midwest Endocrinology Associates, Milwaukee, Wisconsin
  - Cardiovascular Research and Education Foundation, Inc, Wausau, Wisconsin
- Argentina (25):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Concepcion Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Paraná, Entre Ríos Province
  - Novartis Investigative Site, Formosa, Formosa Province
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Grandero Baigorria, Santa Fe Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel, Tucumán Province
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
- Australia (13):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Concord, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Sippy Downs, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Leabrook, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Malvern East, Victoria
  - Novartis Investigative Site, Joondalup, Western Australia
- Austria (4):
  - Novartis Investigative Site, Braunau am Inn
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Hasselt, Limburg
  - Novartis Investigative Site, Aalst, Oost Vlaanderen
  - Novartis Investigative Site, Dendermonde
  - Novartis Investigative Site, Mechelen
- Brazil (22):
  - Novartis Investigative Site, Maceió, Alagoas
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Canoas, Rio Grande do Sul
  - Novartis Investigative Site, Pelotas, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Aracaju, Sergipe
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
  - Novartis Investigative Site, São José dos Campos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Votuporanga, São Paulo
  - Novartis Investigative Site, Campinas
  - Novartis Investigative Site, Rio de Janeiro
- Bulgaria (13):
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Burgas, Burgas
  - Novartis Investigative Site, Blagoevgrad
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Kyustendil
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sandanski
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Varna
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (28):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Red Deer, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, New Minas, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Guelph, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Napean, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Thornhill, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
  - Novartis Investigative Site, Victoriaville, Quebec
- China (37):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Cangzhou, Hebei
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Tangshan, Hebei
  - Novartis Investigative Site, Xingtai, Hebei
  - Novartis Investigative Site, Daqing, Heilongjiang
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Luoyang, Henan
  - Novartis Investigative Site, Pingdingshan, Henan
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Huangshi, Hubei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Changzhou, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Tonghua, Jilin
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Jinzhou, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Xianyang, Shaanxi
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Jining, Shandong
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Zibo, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Lishui, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jining
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (13):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla, Colombia
  - Novartis Investigative Site, Chía, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Ibagué, Tolima Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Manizales
  - Novartis Investigative Site, Medellín
  - Novartis Investigative Site, San Gil
- Croatia (12):
  - Novartis Investigative Site, Zagreb, City of Zagreb
  - Novartis Investigative Site, Osijek, County of Osijek-Baranja
  - Novartis Investigative Site, Krapinske Toplice, Croatia
  - Novartis Investigative Site, Slavonski Brod, Croatia
  - Novartis Investigative Site, Zagreb, Croatia
  - Novartis Investigative Site, Rijeka, Primorje-Gorski Kotar County
  - Novartis Investigative Site, Opatija
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Pula
  - Novartis Investigative Site, Varaždin
  - Novartis Investigative Site, Vinkovci
  - Novartis Investigative Site, Zagreb
- Czechia (27):
  - Novartis Investigative Site, Chlumec nad Cidlinou, Chlumec Nad Cidlinou
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Ostrava, CZE
  - Novartis Investigative Site, Přerov, Olomoucký kraj
  - Novartis Investigative Site, Ostrava, Zabreh
  - Novartis Investigative Site, Brandýs nad Labem
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Český Krumlov
  - Novartis Investigative Site, Hlučín
  - Novartis Investigative Site, Hodonín
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Liberec
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Náchod
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Plzen Bory
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Trutnov
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Ústí nad Labem
  - Novartis Investigative Site, Zlín
  - Novartis Investigative Site, Znojmo
- Denmark (10):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Copenhagen S
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Gandrup
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Herning
  - Novartis Investigative Site, Kobenhavn N V
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Vejle
- Estonia (4):
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Pärnu
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (22):
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valenciennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villeneuve-d'Ascq
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion Crete.
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Thessaloniki
- Hong Kong (4):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Shatin
- Hungary (12):
  - Novartis Investigative Site, Budapest, Pest County
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Hatvan
  - Novartis Investigative Site, Hosszúhetény
  - Novartis Investigative Site, Mosanmagyarovar
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szekszárd
- India (26):
  - Novartis Investigative Site, Guntur, Andhrapradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ajmer, Rajasthan
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Kanpur, Uttar Pradesh
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, Dehradun, Uttrakhand
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Coimbatore
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Uttarakhand
- Israel (10):
  - Novartis Investigative Site, Holon, Gush Dan
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Poria – Neve Oved
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Tel Aviv
- Italy (20):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Caserta, CE
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Chiavari, GE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Latina, LT
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Cinisello Balsamo, MI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Catanzaro
  - Novartis Investigative Site, Napoli
- Latvia (5):
  - Novartis Investigative Site, Liepāja, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Kuldīga
  - Novartis Investigative Site, Ogre
  - Novartis Investigative Site, Riga
- Lithuania (7):
  - Novartis Investigative Site, Kaunas, Kaunas County
  - Novartis Investigative Site, Klaipėda, Klaipėda County
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Panevezys
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Malaysia (13):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Seremban, Negeri Sembilan
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Seri Manjung, Perak
  - Novartis Investigative Site, Taiping, Perak
  - Novartis Investigative Site, Timur Laut, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Miri, Sarawak
  - Novartis Investigative Site, Sungai Buloh, Selangor
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (18):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Actopan, Hidalgo
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Gustavo Adolfo Madero, Mexico City
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Cuernavaca, Morelos
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Tampico, Tamaulipas
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Distrito Federal
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Mexico D F
  - Novartis Investigative Site, Oaxaca City
  - Novartis Investigative Site, Veracruz
- Netherlands (21):
  - Novartis Investigative Site, Arnhem, Gelderland
  - Novartis Investigative Site, Doetinchem, Gelderland
  - Novartis Investigative Site, Nijmegen, Gelderland
  - Novartis Investigative Site, Nijmegen, Gerlderland
  - Novartis Investigative Site, 's-Hertogenbosch, North Brabant
  - Novartis Investigative Site, Tilburg, North Brabant
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Beverwijk, North Holland
  - Novartis Investigative Site, Deventer, Overijssel
  - Novartis Investigative Site, Leeuwarden, Provincie Friesland
  - Novartis Investigative Site, Sneek, Provincie Friesland
  - Novartis Investigative Site, Delft, South Holland
  - Novartis Investigative Site, Dirksland, South Holland
  - Novartis Investigative Site, Dordrecht, South Holland
  - Novartis Investigative Site, The Hague, South Holland
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Venlo
- Philippines (5):
  - Novartis Investigative Site, Iloilo City, Iloilo
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon
  - Novartis Investigative Site, San Juan City
- Poland (19):
  - Novartis Investigative Site, Krakow, Maloposkie
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bygdoszcz
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Grudziądz
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Myszków
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Piotrkow Trybunalski
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (9):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Carnaxide
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Santa Maria da Feira
  - Novartis Investigative Site, Setúbal
  - Novartis Investigative Site, Vila Nova de Gaia
- Research and Cardiovascular Corp, Ponce, Puerto Rico
- Romania (17):
  - Novartis Investigative Site, Piteşti, Argeş
  - Novartis Investigative Site, Oradea, Bihor County
  - Novartis Investigative Site, Buzău, Buzău
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Târgovişte, Dâmbovița County
  - Novartis Investigative Site, Afumaţi, Ilfov
  - Novartis Investigative Site, Baia Mare, Maramureş
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Suceava, Suceava
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Brăila
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Târgu Mureş
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- Slovakia (17):
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Dolný Kubín
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Kráľovský Chlmec
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Ľubochňa
  - Novartis Investigative Site, Malacky
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Rožňava
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Šamorín
  - Novartis Investigative Site, Trnava
- South Africa (10):
  - Novartis Investigative Site, Port Elizabeth, Eastern Cape
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, KwaDukuza, KwaZulu-Natal
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Somerset West, Western Cape
  - Novartis Investigative Site, Cape Town, ZAF
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Western Cape
- Spain (52):
  - Novartis Investigative Site, Ferrol, A Coruna
  - Novartis Investigative Site, Santiago, A Coruna
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Palma, Balearic Islands
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Centelles, Barcelona
  - Novartis Investigative Site, el Prat de Llobregat, Barcelona
  - Novartis Investigative Site, La Roca del Vallès, Barcelona
  - Novartis Investigative Site, Mataró, Barcelona
  - Novartis Investigative Site, Sant Adrià de Besòs, Barcelona
  - Novartis Investigative Site, Vic, Barcelona
  - Novartis Investigative Site, Puerto Real, Cadiz
  - Novartis Investigative Site, Sanlucar Barrameda, Cadiz
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Peralada, Girona
  - Novartis Investigative Site, Las Palmas de Gran C, Las Palmas
  - Novartis Investigative Site, Boadilla del Monte, Madrid
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Antequera, Malaga
  - Novartis Investigative Site, Ronda, Malaga
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Castilleja de la Cuesta, Sevilla
  - Novartis Investigative Site, Lebrija, Sevilla
  - Novartis Investigative Site, Utrera, Sevilla
  - Novartis Investigative Site, Reus, Tarragona
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Almería
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Huelva
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Tarragona
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Sweden (7):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Solna
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Västerås
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Lugano
- Taiwan (7):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (5):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (15):
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Izmir, Bayrakli
  - Novartis Investigative Site, Ankara, Bilkent-Cankaya
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Kadikoy
  - Novartis Investigative Site, Denizli, Kinikli
  - Novartis Investigative Site, Istanbul, Kucukcekmece
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Muğla, Mentese
  - Novartis Investigative Site, Eskişehir, Odunpazari
  - Novartis Investigative Site, Gaziantep, Sehitkamil
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Mersin, Yenisehir
  - Novartis Investigative Site, Istanbul, Zeytinburnu
  - Novartis Investigative Site, Izmir
- United Kingdom (43):
  - Novartis Investigative Site, Luton, Beds
  - Novartis Investigative Site, High Wycombe, Buckinghamshire
  - Novartis Investigative Site, Peterborough, Cambridgeshire
  - Novartis Investigative Site, Connor Downs, Cornwall
  - Novartis Investigative Site, Fowey, Cornwall
  - Novartis Investigative Site, Liskeard, Cornwall
  - Novartis Investigative Site, Newquay, Cornwall
  - Novartis Investigative Site, Exeter, Devon
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Harrow, Middlesex
  - Novartis Investigative Site, Corby, Northamptonshire
  - Novartis Investigative Site, Portadown, Nothern Ireland
  - Novartis Investigative Site, Wansford, Peterborough
  - Novartis Investigative Site, Bristol, South Gloucestershire
  - Novartis Investigative Site, Hardwick, Stockton on Tees
  - Novartis Investigative Site, Bury St Edmunds, Suffolk
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Denbighshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Kettering
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Londonderry
  - Novartis Investigative Site, Middlesex
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Plympton
  - Novartis Investigative Site, Rhyl
  - Novartis Investigative Site, Salford
  - Novartis Investigative Site, Scunthorpe
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Tyne and Wear
  - Novartis Investigative Site, Wiltshire
  - Novartis Investigative Site, Wirrel
  - Novartis Investigative Site, Wrexham
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com